CLINICAL TRIAL: NCT05366465
Title: Specificities of Quality of Life and Influence of Participation on the Quality of Life of the Adult with Spinal Muscular Atrophy in France: a Cross-sectional Study
Brief Title: Quality of Life and Participation of the Adult with Spinal Muscular Atrophy in France
Acronym: QOLSMA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0200
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SMA adult patients
  Interventions: Other: SMA adult patients

INTERVENTIONS:
Other: SMA adult patients — An online questionnaire aimed at collecting demographic and social data, and data concerning activity limitations, participation and quality of life of SMA patients from validated scales : QOLNMD, Rosenberg.

SUMMARY:
Spinal muscular atrophy is a hereditary motorneuron disease caused by a mutation of the SMN1 gene, which is at the origin of a progressive limb and axial motor deficiency. It concerns 1200 individuals in France, including 700 adults in 2018. The main objective of this study is to assess the quality of life of SMA patients in France.

The secondary objectives are, in one hand, to compare the quality of life of SMA patients to a population of neuromuscular diseases patients. And on the other hand to evaluate the determinants of participation and the impact of participation on quality of life in adult SMA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SMA type 1, 2, 3 or 4
* ≥ 18 years old
* giving informed consent to participate to the study
* patients from the study of Dany et al "Construction of a Quality of Life Questionnaire for slowly progressive neuromuscular disease" (2015)

Exclusion Criteria:

* patients who do not complete ≥ 80% of the questionnaire)-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with spinal muscular atrophy in France. And adult NMD patients from the study of Dany et al "Construction of a Quality of Life Questionnaire for slowly progressive neuromuscular disease" (2015)
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
Quality of life | At inclusion
  Quality of life of adult patients with spinal muscular atrophy in France, assessed using the QOLNMD score

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service L'Escale - Médecine Physique et de Réadaptation Pédiatrique Groupement Hospitalier Est des Hospices Civils de Lyon, Bron, Bron
  - VUILLEROT Carole, Bron, Bron

IPD SHARING:
Plan to Share IPD: No